CLINICAL TRIAL: NCT06997263
Title: Comparison Between Two Different Doses of Sublingual Melatonin to Alleviate Anxiety and Pain Associated With Elective Gynecological Surgeries Under General Anesthesia: A Randomized Controlled Trial
Brief Title: Sublingual Melatonin for Anxiety and Pain in Elective Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mariam AbdAllah Ahmed, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS 25-03-2025
Record Dates: First submitted 2024-12-30; First posted 2025-05-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Postoperative Pain; Anesthesia
Keywords: Melatonin; Sublingual Melatonin; Hysterectomy; Ovarian Cystectomy; Myomectomy; Anxiety Reduction; Pain Management; Premedication
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Agnosia | interventions — Melatonin; Administration, Sublingual

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who will collect postoperative anxiety and pain data will be blinded to group assignments to minimize assessment bias. Participants, care providers, and investigators will not be blinded due to the nature of the intervention and its method of administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low-Dose Melatonin Group (Experimental): Participants in this group will receive 3 mg of sublingual melatonin the night before surgery and another 3 mg 1 hour before induction of general anesthesia.
  Interventions: Drug: Melatonin 3 mg Sublingual
- High-Dose Melatonin Group (Experimental): Participants in this group will receive 6 mg of sublingual melatonin the night before surgery and another 6 mg 1 hour before induction of general anesthesia.
  Interventions: Drug: Melatonin 6 mg Sublingual
- Control Grou (No Intervention): Participants in this group will receive no premedication with anxiolytic drugs prior to surgery.

INTERVENTIONS:
Drug: Melatonin 3 mg Sublingual — A single 3 mg dose of sublingual melatonin will be administered the night before surgery and repeated 1 hour before anesthesia induction in participants randomized to the Low-Dose Melatonin Group.
  Arms: Low-Dose Melatonin Group
Drug: Melatonin 6 mg Sublingual — A single 6 mg dose of sublingual melatonin will be administered the night before surgery and repeated 1 hour before anesthesia induction in participants randomized to the High-Dose Melatonin Group.
  Arms: High-Dose Melatonin Group

SUMMARY:
This prospective randomized controlled study aims to evaluate the anxiolytic effect of preoperative sublingual melatonin and its impact on postoperative pain scores when administered in two different doses to female patients undergoing elective gynecological surgeries.

DETAILED DESCRIPTION:
Elective gynecological surgery plays a vital role in women's healthcare, addressing a wide range of medical conditions from benign disorders to oncological diseases. Despite its importance, these procedures often lead to significant preoperative anxiety and postoperative pain, which can adversely affect patient recovery and satisfaction. The psychological impact is particularly prominent in gynecologic surgeries due to factors such as loss of fertility, body image concerns, and invasiveness of the procedures.

The perioperative period is a time of heightened vulnerability, with anxiety potentially leading to physiological stress responses that may compromise surgical outcomes and increase morbidity. Common sources of this anxiety include fear of anesthesia, postoperative pain, surgical failure, and loss of personal control.

To address these concerns, various pharmacologic agents such as benzodiazepines, non-steroidal anti-inflammatory drugs, and opioids have been used. However, these drugs may have limitations or side effects. Recently, melatonin, a naturally occurring hormone involved in regulating the sleep-wake cycle, has been proposed as a promising alternative due to its anxiolytic and analgesic effects. It is considered safe, well-tolerated, and easy to administer.

Sublingual melatonin offers advantages such as rapid absorption and good bioavailability, making it a practical option for preoperative use. This study will explore the comparative efficacy of two different sublingual doses of melatonin on reducing anxiety and postoperative pain in women undergoing elective gynecologic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patient scheduled for open elective gynecological surgeries (hysterectomy, ovarian cystectomy, myomectomy)
* Age 18-65 y
* American Society of Anesthesiologists (ASA) physical status (ASA I -II)

Exclusion Criteria:

* Patients with a history of uncontrolled hypertension
* Ischemic heart disease
* Uncontrolled diabetes
* Bronchial asthma
* Psychiatric illness
* Sleep disorders
* Obesity (Body mass index >30 kg/m2)
* Patients taking antipsychotic, antidepressants, sedatives, anxiolytics, and anti-epileptic drugs.
* Pregnant and lactating females .

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Preoperative Anxiety Score (BAI) | At baseline (preoperative), at recovery (0 hours), and at 12 hours postoperatively
  Anxiety will be assessed using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire. Each item is rated on a 4-point Likert scale (0-3), with total scores ranging from 0 to 63. Higher scores indicate more severe anxiety.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | At 0, 1, 4, 12, and 24 hours postoperatively
  Pain will be assessed using the Numerical Rating Scale (NRS), an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Patients will verbally rate their pain at multiple postoperative time points.
Time to First Rescue Analgesia Request | Up to 24 hours postoperatively
  Duration of postoperative analgesia will be measured as the time from Post-Anesthesia Care Unit (PACU) recovery to the first request for rescue analgesia (morphine), indicating when pain relief wears off.
Cumulative Postoperative Opioid Consumption | From Post-Anesthesia Care Unit (PACU) admission to 24 hours postoperatively
  The total dose of intravenous morphine (mg) administered within the first 24 hours post-surgery to manage postoperative pain.
Post-Anesthesia Care Unit (PACU) Discharge Time | Immediately postoperatively, assessed up to 2 hours
  Time from surgery completion until the patient achieves an Aldrete Recovery Score ≥8, which qualifies them for discharge from Post-Anesthesia Care Unit (PACU). The score assesses activity, respiration, circulation, consciousness, and oxygen saturation (max score = 10).
Length of Hospital Stay | From end of surgery to hospital discharge, typically 1-3 days
  Total time the patient remains hospitalized post-surgery until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Qualiobia, Egypt